CLINICAL TRIAL: NCT00332943
Title: MR Colonography With Fecal Tagging. Barium vs. BariumFerumoxsil
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Collaborators: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: KA-20060039 MA; KA-20060039.
Record Dates: First submitted 2006-06-01; First posted 2006-06-02 (Estimated); Last update posted 2007-09-20 (Estimated); Status verified 2007-09

CONDITIONS: Colorectal Cancer; Polyps
Keywords: colorectal polyps; colorectal cancer; Virtual colonoscopy; Fecal tagging; MR colonography
MeSH Terms: conditions — Colorectal Neoplasms; Polyps

INTERVENTIONS:
Procedure: MR colonography with fecal tagging

SUMMARY:
The purpose of this study is to determine whether Barium or BariumFerumoxsil is better for fecal tagging in MR colonography. Patients referred to colonoscopy are offered MR colonography before colonoscopy. Two days before colonography, patients ingest either a contrast agent A (200 ml Barium sulphate solution 1g/ml)) four times a day or a 200 ml contrast agent B (Barium sulfate(25%) and Ferumoxil(75%)) four times a day, which will render fecal masses "invisible" on the following MR colonography. The patients are randomised to either contrast agent A or B. The examinations are evaluated by two independent blinded readers, who will rate the tagging quality of the contrast agents. The quality of tagging will be rated by a Visual Analog Scale (VAS) and Relative contrast (ReCon = Iwall - Ilumen/ Iwall + Ilumen).

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of colorectal polyps or cancer
* Referred for colonoscopy

Exclusion Criteria:

* Suspicion of IBD
* Pacemaker
* Metal in the body
* Claustrophobia
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-12; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Quality of fecal tagging agent
Sensitivity of VAS score vs. ReCon score

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Achiam, MD, Principal Investigator — Department of Radiology Copenhagen University Hospital Herlev
Locations (1):
- Department of Radiology Copenhagen University Hospital Herlev, Copenhagen, Denmark